CLINICAL TRIAL: NCT01284595
Title: [14C] AZD8931 - A Phase I, Open Label Study of the Absorption, Metabolism, Excretion, and Pharmacokinetics Following a Single Oral Dose to Healthy Male Subjects
Brief Title: Healthy Volunteers, Absorption, Distribution, Metabolism and Excretion (ADME) Study With Single Oral Administration of [14C] AZD8931
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: D0102C00007
Record Dates: First submitted 2011-01-26; First posted 2011-01-27 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
Keywords: Radioactive carbon; Absorption; Distribution; Metabolism; Excretion; Healthy Volunteers
MeSH Terms: interventions — AZD 8931

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZD8931 (Experimental): [14C] AZD8931
  Interventions: Drug: [14C] AZD8931

INTERVENTIONS:
Drug: [14C] AZD8931 — Single 160 mg oral dose administered on Day 1

SUMMARY:
Study to Assess the Absorption, Metabolism and Excretion of [14C]AZD8931 after a Single-Dose Oral Administration

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) of ≥19 and ≤30 kg/m2 and weight of ≥50 kg and ≤100 kg.
* Regular daily bowel movements (ie, production of at least 1 stool per day).
* Non-smokers or ex-smokers who have stopped smoking for >3 months before Visit 1 and have not used nicotine products for >3 months
* Healthy Male volunteers aged 50 to 65 years, inclusive

Exclusion Criteria:

* Healthy volunteers who have been exposed to radiation levels above background (eg, through X-ray examination) of >5 mSv in the last year, >10 mSv in the last 5 years, or a cumulative total of >1 mSv per year of life
* Participation in any prior radiolabelled study within 12 months of the screening visit (Visit 1).
* History of alcohol abuse or excessive intake of alcohol defined as regular weekly intake of 28 units of alcohol or more (1 unit=25 mL spirits, 125 mL wine, 250 mL beer or lager)

Ages: 50 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To investigate the absorption, distribution, metabolism and excretion of AZD931 in human subjects | Multiple blood , urine and faecal samples from pre-dose until 240 hours post last dose
To investigate the pharmacokinetic variable of AZD8931 in plasma | Multiple PK blood samples from pre-dose until 240 hours post last dose

SECONDARY OUTCOMES:
To investigate the safety and tolerability of AZD8931 given orally | Frequent safety measurements during the study from screening period to follow-up
To investigate the AZD8931 metabolites variables in plasma | Multiple PK blood samples from pre-dose until 240 hours post last dose

CONTACTS AND LOCATIONS:
Overall Officials: Darren Wilbraham, MBBS, DCPSA, Principal Investigator — Quintiles Drug Research Unit at Guy's Hospital; Mary Stuart, Study Director — AstraZeneca
Locations (1):
- Research Site, London, United Kingdom

REFERENCES:
- [Derived] Ballard P, Swaisland HC, Malone MD, Sarda S, Ghiorghiu S, Wilbraham D. Metabolic disposition of AZD8931, an oral equipotent inhibitor of EGFR, HER2 and HER3 signalling, in rat, dog and man. Xenobiotica. 2014 Dec;44(12):1083-98. doi: 10.3109/00498254.2014.938257. Epub 2014 Jul 9. PMID 25007130
- See also: Clinical_Study_Protocol_redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1626&filename=D0102C00007_Clinical_Study_Protocol_redacted_for_posting.pdf